CLINICAL TRIAL: NCT04381442
Title: Consequence of Two Protocols and Energy Doses of Low Level Laser Therapy on the Rate of Orthodontic Canine Retraction: A Prospective Clinical Evaluation
Brief Title: Effect of Low Level Laser on Orthodontic Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdullah Mohammed Yahya Al-Haj, Postgraduate MSc. Student, Department of Orthodontics, Faculty of Dental Medicine (Boys), Al-Azhar University, Cairo, Egypt, Dentist, Ministry of Health, Yemen., Al-Azhar University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Laser Effect Canine Movement
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Dental Malocclusion
Keywords: Low Level Laser Therapy; Orthodontic Tooth movement; Canine Retraction; Two Protocols and Energy Doses
MeSH Terms: conditions — Malocclusion | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Buccal &palatal LLLT Group, Buccal &palatal LLLT Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal &palatal low level laser therapy (Experimental): In group I,low level laser therapy was delivered at 10 points; 5 from buccal and 5 from palatal aspects with a total dose of 8 Joule (J) per session that distributed as follows; 2 cervical, 1 middle, 2 apical. Maxillary canines were irradiated with a gallium aluminum-arsenide diode laser in continuous mode with 635 nm, 100 mW, 25 J/cm2, 8 seconds/ point, 0.8 J/point.Maxillary canines were distalized by a standard protocol with uniform 150 gm retraction force via a nickel-titanium closed coil spring.Laser regimen was applied on days 0, 3, 7, and 14 in the 1st month, and thereafter on every 15th day until 6-month observation period of canine retraction phase.
  Interventions: Radiation: Low Level Laser Therapy
- Buccal low level laser therapy (Active Comparator): In group II, low level laser therapy was delivered at 5 points; from buccal palatal aspects only with a total dose of 4 Joule (J) per session that distributed as follows; 2 cervical, 1 middle, 2 apical. Maxillary canines were irradiated with a gallium aluminum-arsenide diode laser in continuous mode with 635 nm, 100 mW, 25 J/cm2, 8 seconds/ point, 0.8 J/point.Maxillary canines were distalized by a standard protocol with uniform 150 gm retraction force via a nickel-titanium closed coil spring.Laser regimen was applied on days 0, 3, 7, and 14 in the 1st month, and thereafter on every 15th day until 6-month observation period of canine retraction phase.
  Interventions: Radiation: Low Level Laser Therapy

INTERVENTIONS:
Radiation: Low Level Laser Therapy
  Other Names: Photobiomodulation

SUMMARY:
The aim of this study was to determine whether orthodontically moved maxillary canines exposed to two different protocols and dosage of LLLT exhibited differences in amount and rate of orthodontic tooth movement.

DETAILED DESCRIPTION:
Fifteen orthodontic patients, 12 females and 3males, with a mean age of 17.48 ± 2.95 years were included. They had a clinical indication for bilateral extraction of at least first maxillary premolars. Using a split mouth design, maxillary left and right sides were randomly divided into two groups. In group 1, LLLT was delivered at 10 points; 5 from buccal and 5 from palatal aspects with a total dose of 8 Joule (J) per session that distributed as follows; 2 cervical, 1 middle, 2 apical. In group II, laser was applied from buccal side only at 5 points through the same order with a dose of 4 J per session. In both protocols, maxillary canines were irradiated with a gallium aluminum-arsenide diode laser in continuous mode with 635 nm, 100 mW, 25 J/cm2, 8 seconds/ point, 0.8 J/point. Both sides were distalized by a standard protocol with uniform 150 gm retraction force via a nickel-titanium closed coil spring. In both protocols, laser regimen was applied on days 0, 3, 7, and 14 in the 1st month, and thereafter on every 15th day until 6-month observation period of canine retraction phase. Amount and monthly rate of maxillary canine retraction and degree of anchorage loss were determined by direct intraoral and indirect 3D digital models measurements. Evaluations were undertaken immediately before initiating retraction (T0), after 4 weeks (T1), after 8 weeks (T2), after 12 weeks (T3), after 16 weeks (T4), after 20 weeks (T5), and after 24 weeks (T6). Significance level was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Complete permanent dentition (3rd molars excluded).
* The age was ranged from 15 -25 years.
* Malocclusion that required extraction of at least maxillary first premolars, followed by canine retraction.
* Good oral hygiene and periodontal health.

Exclusion Criteria:

* Patients who diagnosed to have an indication for non-extraction approach.
* Serious systemic diseases and/or long term medications that could interfere with OTM.
* Previous orthodontic treatment.
* Poor oral hygiene or periodontally compromised patients.
* Craniofacial anomalies or history of parafunctional habits.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Evaluation the rate of maxillary canine retraction | 6 Months
  Evaluation and comparison of amount and monthly rate of distal movement of maxillary canine, in both groups, that were determined by direct intraoral measurements and indirect measurements of 3D scanned study models

SECONDARY OUTCOMES:
Evaluation of anchorage loss | 6 Months
  Evaluation and comparison of the amount of maxillary molar mesial movement (anchorage loss) between both groups via study models assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Al-Haj, MSc student, Principal Investigator — Al-Azhar University; Farouk A Hussein, Ass.Prof, Study Director — Al-Azhar University